CLINICAL TRIAL: NCT02234102
Title: Eagle AF - Endoscopically Guided Laser Ablation of Persistent Atrial Fibrillation
Brief Title: Eagle AF (Atrial Fibrillation) - Endoscopically Guided Laser Ablation of Persistent Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof. Dr. med. Bernd Lemke (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Bernd Lemke, Klinikdirektor der Klinik für Innere Medizin III, Märkische Kliniken GmbH
Organization: Märkische Kliniken GmbH (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF 34/2014 version 02
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paroxysmal Atrial Fibrillation (PAF) (Active Comparator): Endoscopically guided laser ablation
  Interventions: Device: Endoscopically guided laser ablation HeartLight system
- Persistent Atrial Fibrillation (Active Comparator): Endoscopically guided laser ablation
  Interventions: Device: Endoscopically guided laser ablation HeartLight system

INTERVENTIONS:
Device: Endoscopically guided laser ablation HeartLight system
  Other Names: HeartLight system

SUMMARY:
The study aims to compare the results of pulmonary vein isolation (PVI) with a single technology approach in patients suffering from paroxysmal atrial fibrillation (PAF) with patients who have persistent AF of less than 3 months. Many studies have shown that electrical reconnection of the pulmonary veins following the index procedure can occur in up to 40% of targeted veins leading to a recurrence of PAF. Endoscopically guided laser ablation utilising the HeartLight system (CardioFocus Inc., USA) has been shown to be safe and effective and has also shown promising rates of durable isolation compared to point by point radio frequency techniques. However, the impact of employing this technique for patients with persistent AF has not yet been reported. The study hypothesis is that there will be no statistically significant difference between the results of PVI in the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* failure of at least one specific class I or III antiarrhythmic drug (AAD)
* left atrial size < 50 mm
* left ventricular ejection fraction > 45%
* others
* specific for PAF: diagnosed with self-terminating episodes for no longer than 7 days
* specific for persistent AF: diagnosed with episodes of > 7 days and < 90 days

Exclusion Criteria:

* AF secondary to a reversible cause of non-cardiac origin
* uncontrollable hypertension
* left atrial thrombus
* others
* specific for PAF: more than 1 electrical cardioversion in the year prior to enrollment
* specific for persistent AF more than 4 electrical cardioversions in the year prior to enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Documented recurrence of AF or any tachyarrhythmia lasting > 30 seconds | Between day 90 and 365 after index procedure

SECONDARY OUTCOMES:
Number of electrical cardioversions needed | 365 days after index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Lemke, Prof. Dr., Principal Investigator — Klinikum Lüdenscheid Klinik f. Innere Medizin III
Locations (3):
- Germany (3):
  - St.Vinzenz-Hospital GmbH, Cologne, North Rhine-Westphalia
  - Märkische Kliniken GmbH, Klinik für Innere Medizin III, Lüdenscheid, North Rhine-Westphalia
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin, State of Berlin